CLINICAL TRIAL: NCT02673762
Title: Salivary Transcriptome Biomarkers for Early Diabetes Detection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: PeriRx (Industry)
Responsible Party: Sponsor
Other Study IDs: PeriRx003
Record Dates: First submitted 2015-12-19; First posted 2016-02-04 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Pre-diabetes; Type II Diabetes; Insulin Resistance
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Salivary mRNA and cDNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal glucose metabolism: Normal fasting blood glucose, 2 hour post prandial glucose, hemoglobin A1c and HOMA IR
- Pre-diabetes: Abnormal glucose tolerance tests and/or insulin resistance with fating blood glucose and hemoglobin A1c below type II diabetes levels
- Type II diabetes: Hemoglobin A1c 6.5% or greater, fasting blood glucose >125 mg/dl or 2 hour post-prandial blood glucose 200 mg/ml or greater

SUMMARY:
A PRoBE design study will be used to obtain saliva from patients before undergoing blood study evaluation for screening at risk patients for the presence of undiagnosed pre-diabetes of type II diabetes. Pre-specified saliva biomarkers will be evaluated along with multi-marker models for their discriminatory value for distinguishing patients with normal glucose metabolism from those with disease. Appropriate housekeeping genes will also be incorporated to allow for the measurement of relative gene expression.

DETAILED DESCRIPTION:
Prospective-specimen-collection, retrospective-blinded-evaluation (PRoBE) methods will be employed to collect saliva and evaluate transcriptome markers for early pre-diabetes and type II diabetes identification. At risk patients will have fasting blood glucose and insulin levels measured along with hemoglobin A1c and 2 hour post-prandial glucose levels. Saliva samples will be stored and will be analyzed after pre-specifying a panel of mRNAs and a multi marker model for validation. The pre-specified mRNAs and multi-marker model will be determined after analysis of data from a currently ongoing case-control study. After analyzing the data from this prior trial a validation plan will be locked before analysis of the prospectively collected specimens. Pre-diabetes will be defined based on abnormal glucose tolerance tests. Insulin resistance will be calculated as HOMA IR. The diagnostic value of the salivary transcriptome for will be compared with that of hemoglobin A1c and fasting blood glucose for the detection of pre-diabetes, insulin resistance and type II diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with unknown glucose metabolism status and
* Requiring clinically driven screening for abnormal glucose metabolism and
* Outpatient status

Exclusion Criteria:

* Patients on treatment for abnormal glucose metabolism including diet and drug therapy
* Patients with a prior diagnosis of abnormal glucose metabolism
* Patients on treatment with corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with undiagnosed abnormal glucose metabolism undergoing clinically driven screening for pre-diabetes and type II diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
A multi marker test score based on a pre-specified model is measured in each patient. The test score is on a scale of 0 to 1.0 and relates to the probability of disease. | At study entry
  The area under the ROC curve is used to determine the overall performance of the model at the completion of the study. An area over 0.7 is considered clincially significant.

SECONDARY OUTCOMES:
Pre-specified mRNA marker Ct values from PCR analysis will be measured in individual patients | At study entry
  The performance of each individual marker will be determined at study completion my comparing median values between groups by nonparametric analysis. A p value of less than or equal to 0.05 is considered significant.
Housekeeping gene Ct values on PCR analysis will be measured in individual patients | At study entry
  The performance of these genes will be determined based on stability within and between groups utilizing the NormFinder program. Stability values of < 0.2 will be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Jack L Martin, MD, Principal Investigator — San Antonio Endovascular and Heart Institute
Locations (1):
- San Antonio Endovascular and Heart Institute, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No